CLINICAL TRIAL: NCT05221723
Title: Functional Interval Training for People With Spinal Cord Injury and Their Care Partners
Acronym: SCI-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Colleges of Health Education (Other)
Responsible Party: Principal Investigator, Kaci Handlery, Assistant Professor, School of Physical Therapy, Arkansas Colleges of Health Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT-2021-024
Record Dates: First submitted 2022-01-09; First posted 2022-02-03 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; exercise; physical activity
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Group (Experimental): In this single group design, all participants will be provided with 6 months of twice weekly supervised group exercise.
  Interventions: Behavioral: High Intensity Interval Exercise Training Group

INTERVENTIONS:
Behavioral: High Intensity Interval Exercise Training Group — Participants will participate in a maximum of twice weekly exercise classes (90 minutes each class) for a total of 6 months. While participants will be encouraged to attend as many classes as able, there is no minimum requirement for class attendance. During the exercise classes, participants will participate in a 10-minute warm up, followed by 30-60 minutes of aerobic, resistance and/or balance training up to a maximum intensity of 8/10 on the rating of perceived exertion scale. Participants will finish each class with a 10-minute cool-down consisting of lower intensity exercise.

SUMMARY:
Functional Interval Training for People with Spinal Cord Injury and Their Care Partners (SCI-FIT) aims to address barriers to physical activity for people with spinal cord injury and their care partners. This research study provides free, twice weekly group-based, adaptable exercise classes for people with spinal cord injury and their care partners.

DETAILED DESCRIPTION:
Regular physical activity, and more specifically exercise, is beneficial for people with and without spinal cord injury (SCI). Unfortunately, people with spinal cord injury (pSCI) are less physically active than adults without SCI and are at an increased risk of cardiovascular disease. Care partners, or those who provide frequent assistance to those living with SCI, also achieve low physical activity levels and share similar health risks as a result. Often there are limited opportunities for pSCI to engage in regular exercise. In addition, pSCI and their care partners often face significant barriers to exercise including 1) lack of exercise participation opportunities; 2) cost of quality exercise instruction; 3) inaccessible exercise equipment or environments; 4) lack of social support from family and peers. This study, Functional Interval Training for People with Spinal Cord Injury and Their Care Partners (SCI-FIT) will explicitly address the barriers to exercise pSCI and their care partners often face with the primary goals of improving the health, physical activity levels, and quality of life of pSCI and their care partners. In order to address these goals, SCI-FIT will provide no-cost, twice weekly, group-based, adaptable exercise programming for pSCI and their care partners. All participants will be required to have physician or advanced practice provider clearance to exercise and will be evaluated by a physical therapist at no-cost prior to beginning the intervention to assess eligibility for the study. All eligible participants will complete a demographics questionnaire and will undergo a battery of baseline outcome assessments prior to undergoing the exercise intervention. Participants will complete 6-months of twice weekly group exercise classes aimed and hypothesized to increase physical activity levels, muscular strength, social support for exercise, functional mobility, peak power output, aerobic capacity, and quality of life for people with spinal cord injury and their care partners. Participants will repeat baseline outcome assessments at study midpoint (3-months) and study completion (6-months).

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury: Must have a clinical diagnosis of spinal cord injury at level C5 (ASIA A-D) and/or must possess at least 4/5 elbow flexion muscular strength
* Care Partners: self-identified care partner of a person with spinal cord injury participating in the study
* Must be at least 18 years of age
* Must be able to communicate and read in English
* Must have physician or advanced practice provider clearance to exercise
* Must provide their own transportation to and from the research study
* Must be able to ambulate independently and/or propel a power or manual wheelchair independently
* Care Partners: self-identified care partner of a person with spinal cord injury participating in the study

Exclusion Criteria:

* Less than 4/5 elbow flexion muscular strength
* Unable to ambulate independently or propel a power or manual wheelchair independently
* Unable to provide transportation to and from the research study
* Unable to communicate in English
* Unable to present documented medical clearance to exercise from physician or advanced practice provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Participant Attendance | 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  The percentage of interventions sessions attended by participants.

SECONDARY OUTCOMES:
Change in 6-Minute Arm Test (6-MAT) at 6 Months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Assessment of aerobic capacity in individuals with spinal cord injury
Change in Five Times Sit to Stand Test at 6 Months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Participants who are able to stand will complete this assessment of lower extremity strength over three trials.
Change in Upper Extremity Muscular Strength at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Muscular strength of the upper extremities will be assessed via 3-trials of hand-held dynamometry of the shoulder flexor, shoulder extensor, elbow flexor and elbow extensor muscle groups as well as grip strength via a dynamometer.
Change in The Spinal cord Injury Exercise Self-Efficacy Scale at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Measures perceived self-efficacy for various types of physical activities for people with spinal cord injury. The scale has a minimum score of 10 and a maximum score of 40. Higher scores indicate greater confidence in planning and carrying out physical activities and/or exercise based on their own volition.
Change in Self Efficacy for Exercise Scale at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Self report measure for exercise self efficacy completed by care partner participants. The minimum score is 0 and maximum score is 90. A higher score indicates higher self-efficacy for exercise.
Change in Social Support and Exercise Survey at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Self report measure for social support for exercise from family and friends. The scale has a minimum score of 46 and maximum score of 230. Higher scores indicate greater social support of friends and family for physical activity and exercise behaviors.
Change in Gait Speed at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Measure of walking speed at both self-selected and fast walking speed for ambulatory participants.
Change in Rand 36-Item Health Survey 1.0 at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Self-reported measure of health related quality of life for participants who are care partners. The measure assesses eight health concepts through eight subscales (physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions). Scores in each category are averaged and range from 0 to 100, with higher scores indicating better health-related quality of life.
Change in Quality of Life for People with Spinal Cord Injury as assessed by the Spinal Cord Injury - Quality of Life Measure [Emotional Health and Social Participation] at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Self report measure of quality of life related to Emotional Health (positive affect and well-being, resilience, self-esteem, and stigma) and Social Participation (independence) for people with spinal cord injury.
Change in Spinal Cord Injury - Functional Index at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Self report measure of perceived functional abilities of people with spinal cord injury including self-care, basic mobility, ambulation, manual wheelchair, power wheelchair, and ambulation.
Change in One Minute Peak Power Test at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Measure of peak power assessed via a 1-minute skiergometer tests
Change in Moderate to Vigorous Physical Activity Levels at 6 Months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Physical activity levels will be measured via wrist worn Actigraph GT9X Link. The Actigraph is able to detect acceleration in multiple planes of motion. Through collecting acceleration data, different intensities of physical activity will be inferred (i.e light, moderate and vigorous intensity physical activity), with moderate-to-vigorous intensity physical activity being used as the primary outcome measure. At the four time points, participants will wear the Actigraph for 7 consecutive days. The Actigraph will not need to be removed for activities such as bathing and showering, however the device will be removed for activities such as swimming.
Participant Retention | After 6 months of exercise intervention
  The number and percentage of participants who remain in the study through the final measurement point at 6 months.
Change in lower extremity functional strength at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Lower extremity strength will be measured via functional test (Five Times Sit to Stand). This test records the amount of time taken to rise and sit to and from a chair five consecutive times. Faster times indicate greater lower extremity strength.
Change in 6 Minute Walk Test at 6 months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  The 6 Minute Walk Test measures a participants ability to cover as much distance (measured in meters) as possible while walking for 6 minutes. Participants will walk along a pre-defined pathway for 6 minutes, resting as needed. The test is a measure of walking endurance with further distances indicating greater endurance.
Change in Global Rating of Change at 6 Months | After 6 months of exercise intervention
  Participants will rate their perceived level of change on a 15-point Likert Scale ranging from -7 (a very great deal less/worse to +7 (a very great deal more/better) with 0 representing no change. They will use this scale to answer 4 separate questions: 1) amount of physical activity performed in an average week, 2) ability to walk or push leisurely, 3) ability to walk or push fast, 4) ability to walk or push for a long period of time.
Change in Self-Reported Physical Activity Level at 6 Months | Baseline, 3 months (intervention midpoint), 6 months (immediately post intervention completion)
  Participants report their perceived physical activity levels compared to people their own age using a 5-point Likert Scale ranging from "much more active" to "much less active".
Participant Recruitment Rate | Throughout the 6-month study period
  The number of participants recruited will be reported as a percentage of total participants contacted for study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Kaci Handlery, DPT, Principal Investigator — Arkansas Colleges of Health Education
Locations (1):
- Arkansas Colleges of Health Education, Fort Smith, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hol AT, Eng JJ, Miller WC, Sproule S, Krassioukov AV. Reliability and validity of the six-minute arm test for the evaluation of cardiovascular fitness in people with spinal cord injury. Arch Phys Med Rehabil. 2007 Apr;88(4):489-95. doi: 10.1016/j.apmr.2006.12.044. PMID 17398251
- [Background] Murray D, Hardiman O, Campion A, Vance R, Horgan F, Meldrum D. The effects of a home-based arm ergometry exercise programme on physical fitness, fatigue and activity in Polio survivors: a randomised controlled trial. Clin Rehabil. 2017 Jul;31(7):913-925. doi: 10.1177/0269215516661225. Epub 2016 Aug 16. PMID 27530605
- [Background] Totosy de Zepetnek JO, Au JS, Hol AT, Eng JJ, MacDonald MJ. Predicting peak oxygen uptake from submaximal exercise after spinal cord injury. Appl Physiol Nutr Metab. 2016 Jul;41(7):775-81. doi: 10.1139/apnm-2015-0670. Epub 2016 Mar 15. PMID 27363732
- [Background] Tawashy AE, Eng JJ, Krassioukov AV, Miller WC, Sproule S. Aerobic exercise during early rehabilitation for cervical spinal cord injury. Phys Ther. 2010 Mar;90(3):427-37. doi: 10.2522/ptj.20090023. Epub 2010 Jan 21. PMID 20093326
- [Background] Tulsky DS, Kisala PA, Victorson D, Tate DG, Heinemann AW, Charlifue S, Kirshblum SC, Fyffe D, Gershon R, Spungen AM, Bombardier CH, Dyson-Hudson TA, Amtmann D, Kalpakjian CZ, Choi SW, Jette AM, Forchheimer M, Cella D. Overview of the Spinal Cord Injury--Quality of Life (SCI-QOL) measurement system. J Spinal Cord Med. 2015 May;38(3):257-69. doi: 10.1179/2045772315Y.0000000023. PMID 26010962
- [Background] Crane DA, Hoffman JM, Reyes MR. Benefits of an exercise wellness program after spinal cord injury. J Spinal Cord Med. 2017 Mar;40(2):154-158. doi: 10.1179/2045772315Y.0000000038. Epub 2015 Jun 25. PMID 26108561
- [Background] Hicks AL, Martin KA, Ditor DS, Latimer AE, Craven C, Bugaresti J, McCartney N. Long-term exercise training in persons with spinal cord injury: effects on strength, arm ergometry performance and psychological well-being. Spinal Cord. 2003 Jan;41(1):34-43. doi: 10.1038/sj.sc.3101389. PMID 12494319
- [Background] Nash MS. Exercise as a health-promoting activity following spinal cord injury. J Neurol Phys Ther. 2005 Jun;29(2):87-103, 106. doi: 10.1097/01.npt.0000282514.94093.c6. PMID 16386165
- [Background] Post MW, Bloemen J, de Witte LP. Burden of support for partners of persons with spinal cord injuries. Spinal Cord. 2005 May;43(5):311-9. doi: 10.1038/sj.sc.3101704. PMID 15685263
- [Background] Anneken V, Hanssen-Doose A, Hirschfeld S, Scheuer T, Thietje R. Influence of physical exercise on quality of life in individuals with spinal cord injury. Spinal Cord. 2010 May;48(5):393-9. doi: 10.1038/sc.2009.137. Epub 2009 Oct 20. PMID 19841634
- [Background] Lynch J, Cahalan R. The impact of spinal cord injury on the quality of life of primary family caregivers: a literature review. Spinal Cord. 2017 Nov;55(11):964-978. doi: 10.1038/sc.2017.56. Epub 2017 Jun 27. PMID 28653672
- [Background] LaVela SL, Landers K, Etingen B, Karalius VP, Miskevics S. Factors related to caregiving for individuals with spinal cord injury compared to caregiving for individuals with other neurologic conditions. J Spinal Cord Med. 2015 Jul;38(4):505-14. doi: 10.1179/2045772314Y.0000000240. Epub 2014 Jul 3. PMID 24993244